CLINICAL TRIAL: NCT07242612
Title: Determination of Selective Bone Turnover Markers and Their Association With Treatment Efficacy in Primary Postmenopausal Osteoporotic Women: A Randomized Control Trial
Brief Title: Bone Turnover Markers and Treatment Efficacy in Postmenopausal Osteoporosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/008
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal
Keywords: Bone Turnover Markers; Bone Density; Postmenopausal Osteoporosis; DEXA Scan
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Alendronate; Ibandronic Acid; Risedronic Acid; Teriparatide

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel treatment groups to receive different drug interventions concurrently.
Who Masked: Participant, Investigator
Masking Description: The protocol states this will be a "double blinded study" where "the participant and researcher will be unaware of the interventions until the participants complete their 6 months of interventions. Only the research assistant will be aware of the interventions given."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anabolic Therapy Group (Experimental): Participants in this group will receive the anabolic drug Teriparatide 20 mcg, administered as a daily subcutaneous injection, for a duration of 6 months. In addition, all participants in this arm will receive daily Calcium and Vitamin D supplements.
  Interventions: Drug: Teriparatide
- Antiresorptive Therapy Group (Active Comparator): Participants will receive one of the following oral antiresorptive drugs for 6 months: Alendronate 70mg weekly, Ibandronate 150mg monthly, or Risedronate 150mg monthly. All participants will also receive Calcium and Vitamin D supplementation.
  Interventions: Drug: Alendronate, Ibandronate; Risedronate

INTERVENTIONS:
Drug: Alendronate, Ibandronate; Risedronate — Oral bisphosphonate tablets. Participants will receive one of the following specific regimens: Alendronate 70mg taken once per week, Ibandronate 150mg taken once per month, or Risedronate 150mg taken once per month. This is combined with daily Calcium and Vitamin D supplementation. The total treatment duration is 6 months.
  Other Names: Fosamax; Bonviva; Actonel
  Arms: Antiresorptive Therapy Group
Drug: Teriparatide — A solution for subcutaneous injection. The dosage is 20 micrograms (mcg) injected once daily. This is combined with daily Calcium and Vitamin D supplementation. The total treatment duration is 6 months.
  Other Names: Forteo
  Arms: Anabolic Therapy Group

SUMMARY:
This study investigates the use of blood tests known as Bone Turnover Markers (BTMs) to quickly monitor the effectiveness of osteoporosis treatment in postmenopausal women. Osteoporosis, which weakens bones and increases fracture risk, is typically monitored using a DEXA scan to measure bone density (BMD), but this method changes slowly. BTMs may show a response to medication within just 3 to 6 months. In this randomized controlled trial, 40 postmenopausal women with osteoporosis will be assigned to receive either antiresorptive drugs (which slow bone loss) or anabolic drugs (which build new bone), along with calcium and vitamin D. The study will compare how these treatments affect BTMs and BMD over six months to determine if BTMs can serve as an early and reliable indicator of treatment success, which could be particularly useful in regions like Pakistan where access to repeated DEXA scans is limited.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to evaluate the association between selective BTM and the efficacy of different drug therapies in primary postmenopausal osteoporotic women. The study is motivated by the high prevalence of osteoporosis in this demographic in Pakistan and the limitations of the current gold standard, BMD measured by DEXA scan, which reflects changes in bone strength at a delayed rate. BTMs, being biochemical indicators of bone formation and resorption, offer a dynamic and rapid assessment of bone metabolic activity, potentially providing an early measure of treatment response within months rather than years. The trial will enroll 40 eligible women over 50, who will be randomly and blindly assigned to one of two treatment groups: one receiving antiresorptive drugs (such as Alendronate) and the other receiving anabolic drugs (Teriparatide), both supplemented with calcium and vitamin D for a six-month period. The primary outcomes include the comparative change in specific BTMs (BsALP, TRACP-5b, and Sclerostin) at three and six months, and the change in BMD at six months. Secondary outcomes will assess the correlation between BTM and BMD changes, as well as fracture incidence and quality of life. By analyzing these parameters, the study aims to generate valuable evidence for the utility of BTMs in guiding and monitoring osteoporosis treatment in a Pakistani clinical setting, potentially leading to more responsive and personalized patient management.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (at least one year since last menstrual cycle).
* Age greater than 50 years.
* Diagnosis of primary osteoporosis.
* Currently not on any anti-osteoporosis medications.
* Not taking Calcium or Vitamin D supplements.
* Volunteer to participate and provide informed consent.

Exclusion Criteria:

* Women with multiple vertebral fractures or severe lumbar degenerative changes.
* Use of hormone/estrogen therapy, calcitonin, oral bisphosphonates, IV ibandronate, IV Zoledronic acid, denosumab, or teriparatide within the past 18 months.
* Use of corticosteroids (short or long-term).
* History of hyperthyroidism, hypothyroidism, liver disease, kidney disease, or tumors.
* Presence of secondary causes of osteoporosis (e.g., eating disorders, celiac disease, diabetes, hematologic disorders).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Bone Turnover Markers (BTMs) | Baseline, 3 months, and 6 months.
  Mean change from baseline in the serum levels of specific bone turnover markers, including the bone formation marker Bone-Specific Alkaline Phosphatase (BsALP) and the bone resorption marker Tartrate-Resistant Acid Phosphatase 5b (TRACP-5b), and the osteocyte marker Sclerostin.
Change in Bone Mineral Density (BMD) | Baseline and 6 months.
  Mean change from baseline in Bone Mineral Density (BMD) T-score as measured by Dual-Energy X-ray Absorptiometry (DEXA) scans at the hip, spine, and femoral neck.

SECONDARY OUTCOMES:
Incidence of New Fractures | Through study completion, an average of 6 months.
  The number of participants who experience any new fragility fractures during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Mehmood, PhD Scholar, Principal Investigator — Institute of Basic Medical Sciences, Khyber Medical University; Rubina Nazli, PhD, Study Director — Institute of Basic Medical Sciences, Khyber Medical University; Arshad Hussain, M.D Consultant, Principal Investigator — Northwest General Hospital, Peshawar; Ehtesham Khan, PhD, Principal Investigator — InsInstitute of Basic Medical Sciences, Khyber Medical University
Locations (1):
- Northwest General Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
A definitive plan for sharing individual participant data has not been established. The data collected, including de-identified individual participant records for primary and secondary outcomes, may be made available upon reasonable request after the primary results are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data may become available beginning 6 months after the publication of the primary study findings and will be accessible for a period of 3 years.
Access Criteria: Access to IPD will be considered for researchers who provide a methodologically sound proposal. Requests should be directed to the corresponding author. Approval will be subject to review by the study's supervisory committee and a signed data sharing agreement.

REFERENCES:
- [Background] Lorentzon M, Branco J, Brandi ML, Bruyere O, Chapurlat R, Cooper C, Cortet B, Diez-Perez A, Ferrari S, Gasparik A, Herrmann M, Jorgensen NR, Kanis J, Kaufman JM, Laslop A, Locquet M, Matijevic R, McCloskey E, Minisola S, Pikner R, Reginster JY, Rizzoli R, Szulc P, Vlaskovska M, Cavalier E. Algorithm for the Use of Biochemical Markers of Bone Turnover in the Diagnosis, Assessment and Follow-Up of Treatment for Osteoporosis. Adv Ther. 2019 Oct;36(10):2811-2824. doi: 10.1007/s12325-019-01063-9. Epub 2019 Aug 22. PMID 31440982
- [Background] Bhattoa HP, Cavalier E, Eastell R, Heijboer AC, Jorgensen NR, Makris K, Ulmer CZ, Kanis JA, Cooper C, Silverman SL, Vasikaran SD; IFCC-IOF Committee for Bone Metabolism. Analytical considerations and plans to standardize or harmonize assays for the reference bone turnover markers PINP and beta-CTX in blood. Clin Chim Acta. 2021 Apr;515:16-20. doi: 10.1016/j.cca.2020.12.023. Epub 2020 Dec 28. PMID 33382995
- [Background] Nadeem S, Pervez A, Abid MA, Khalid RN, Rizvi NA, Aamdani SS, Ayub B, Mustafa MA, Ahmed S, Riaz M, Irfan K, Noordin S, Jafri L, Majid H, Umer M, Zehra N, Sheikh A, Haider AH, Khan AH. GRADE-ADOLOPMENT of clinical practice guideline for postmenopausal osteoporosis management-a Pakistani context. Arch Osteoporos. 2023 May 19;18(1):71. doi: 10.1007/s11657-023-01258-2. PMID 37204537
- [Background] Jorgensen NR, Mollehave LT, Hansen YBL, Quardon N, Lylloff L, Linneberg A. Comparison of two automated assays of BTM (CTX and P1NP) and reference intervals in a Danish population. Osteoporos Int. 2017 Jul;28(7):2103-2113. doi: 10.1007/s00198-017-4026-z. Epub 2017 Apr 28. PMID 28455749
- [Background] Moller AMJ, Delaisse JM, Olesen JB, Canto LM, Rogatto SR, Madsen JS, Soe K. Fusion Potential of Human Osteoclasts In Vitro Reflects Age, Menopause, and In Vivo Bone Resorption Levels of Their Donors-A Possible Involvement of DC-STAMP. Int J Mol Sci. 2020 Sep 2;21(17):6368. doi: 10.3390/ijms21176368. PMID 32887359
- [Background] Patel D, Worley JR, Volgas DA, Crist BD. The Effectiveness of Osteoporosis Screening and Treatment in the Midwest. Geriatr Orthop Surg Rehabil. 2018 Mar 29;9:2151459318765844. doi: 10.1177/2151459318765844. eCollection 2018. PMID 29623238
- [Background] Rizzoli R. Postmenopausal osteoporosis: Assessment and management. Best Pract Res Clin Endocrinol Metab. 2018 Oct;32(5):739-757. doi: 10.1016/j.beem.2018.09.005. Epub 2018 Sep 22. PMID 30449552
- [Background] Cosman F, McMahon D, Dempster D, Nieves JW. Standard Versus Cyclic Teriparatide and Denosumab Treatment for Osteoporosis: A Randomized Trial. J Bone Miner Res. 2020 Feb;35(2):219-225. doi: 10.1002/jbmr.3850. Epub 2019 Oct 23. PMID 31419313